CLINICAL TRIAL: NCT00374556
Title: The Efficacy of Eszopiclone (Lunesta) for Chronic Insomnia Associated With Osteoarthritis.
Brief Title: Insomnia and Osteoarthritis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00001703
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Insomnia
Keywords: eszopiclone; insomnia
MeSH Terms: conditions — Osteoarthritis; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Eszopiclone (Experimental): Eszopiclone 3mg capsules, once daily at bedtime for 12 weeks
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): 3mg placebo capsule, once daily at bedtime for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 3mg placebo capsule, once daily at bedtime
  Arms: Placebo
Drug: Eszopiclone — 3mg capsule, once daily at bedtime
  Arms: Eszopiclone

SUMMARY:
This research is being done to evaluate the effects of a sleeping pill (eszopiclone, Lunesta)in patients with arthritis of the knee who also suffer from chronic insomnia. This study will test whether Lunesta improves sleep, pain sensitivity, and daytime symptoms in patients with knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Diagnosed with and under physicians care for osteoarthritis of the knee according to American College of Rheumatology Criteria with radiographic evidence demonstrating at least grade 1 osteoarthritis (OA)
* Report at least typical arthritic pain>4 out of 10 (0=no pain, 10=the most extreme pain imaginable)
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and International Classification of Sleep Disorders, Revised definition (ICSD-R) criteria for either primary (psychophysiologic) insomnia or insomnia secondary to osteoarthritis
* Insomnia symptoms must include problems with middle of the night awakenings
* Insomnia symptom duration > 6 months
* Baseline, 2-week, sleep diary average wake after sleep onset time >30 minutes
* Baseline self-reported total sleep time < 6.5 hours per night
* Patients taking NSAID therapy for pain must be on a stable dose for a period of at least one month prior to initiating the study

Exclusion Criteria:

* Intrinsic sleep disorders other than insomnia (sleep apnea, periodic limb movement disorder, etc)
* Significant rheumatologic or chronic pain disorders other than osteoarthritis of the knee, including fibromyalgia or the complaint of widespread pain impacting 4 quadrants, complex regional pain syndrome, post herpetic neuralgia, etc)
* Major medical disease (including, hepatic impairment, chronic obstructive pulmonary disease/compromised respiratory function, cancer, dementia, diabetes, congestive heart failure, cerebrovascular disease, raynaud's syndrome)
* Active major psychiatric disorders (including dementia or cognitive impairment) and history of schizophrenia or bipolar I disorder
* History of serious suicide attempt; 6) history of alcohol or substance (including prescription medications) abuse
* Pregnancy or plans to become pregnant within 6 months
* Intraarticular steroid injection within the past month
* Regular (>3 days/week) use of antidepressants, antipsychotics, and mood stabilizers, within the past two months
* Regular (> 3/week) use of myorelaxants, narcotics, sedative hypnotics, and anticonvulsants within the past one month
* Unwilling or unable to discontinue all use of the medications listed in #10 for two weeks prior to starting the study
* Unwilling or unable to discontinue all centrally acting agents and all analgesic usage within 24 hours of pain testing sessions
* Refusal to provide consent to contact patient's physician to establish diagnosis and obtain medical record information
* Regular tobacco or nicotine use
* Heavy caffeine use [(>2 cups of coffee/day (equivalent)
* History of previous allergic reaction or severe side effects to sedative hypnotics
* Use of potent CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, troleandomycin, ritonavir, nelfinavir)
* In addition, subjects will undergo in-laboratory blood tests prior to receiving drug and will be excluded from further participation if they exhibit: a) positive pregnancy test, b) positive toxicology (benzodiazepine, opioids, Tetrahydrocannabinol (THC), alcohol, and stimulants), c) abnormal liver enzyme panel

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Smith, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 were assessed for eligibility. 75 were excluded based on not meeting inclusion criteria. 30 were randomized to one of 2 arms. One subject after randomization ( to placebo condition) was determined to be ineligible due to failing sleep apnea entry criteria. They were removed from the study and did not contribute to baseline data.
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 14 | 16
Completed | 13 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Removed at baseline due to medical cond | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only calculated for the 29 participants above. One subject after randomization ( to placebo condition) was determined to be ineligible due to failing sleep apnea entry criteria. They were removed from the study and did not contribute to baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.64 (5.18) | 52.93 (6.64) | 53.76 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
Kellgren Lawrence OA grade [Mean (Standard Deviation); unit: units on a scale] — grade 0: no radiographic features of osteoarthritis (OA) are present grade 1: doubtful joint space narrowing (JSN) and possible osteophytic lipping grade 2: definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph grade 3: multiple osteophytes, definite JSN, sclerosis, possible bony deformity grade 4: large osteophytes, marked JSN, severe sclerosis and definite bony deformity
  units on a scale
    Right knee | 2.08 (0.86) | 1.53 (0.91) | 1.79 (0.92)
    Left Knee | 2.07 (1.07) | 1.79 (1.05) | 1.93 (1.05)
Kellgren Lawrence OA grade >=3 in either knee [Number; unit: participants] — grade 0: no radiographic features of OA are present grade 1: doubtful joint space narrowing (JSN) and possible osteophytic lipping grade 2: definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph grade 3: multiple osteophytes, definite JSN, sclerosis, possible bony deformity grade 4: large osteophytes, marked JSN, severe sclerosis and definite bony deformity
  participants | 6 | 4 | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.41 (5.21) | 31.36 (6.53) | 30.42 (5.91)
Duration of OA [Mean (Standard Deviation); unit: months] | 87.7 (98.06) | 108.5 (95.11) | 95.6 (95.69)

OUTCOME MEASURES:

1. Primary Outcome: Wake After Sleep Onset (WASO)
Description: Total minutes of wakefulness recorded after sleep onset. (Recorded in Daily Sleep Diary) WASO= time awake in the middle of the night, not counting SL or time in bed after awakening. Recorded in minutes
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: Data was not included for all participants, as some were unable to complete the task or experienced technical difficulties.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
minutes
  Baseline | 117.33 (108.09) | 88.0 (57.26)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 81.00 (98.76) | 65.56 (67.28)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 61.94 (55.59) | 58.57 (51.85)

2. Primary Outcome: Time in Bed
Description: Total time in bed, in minutes
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
minutes
  Baseline | 464.00 (134.31) | 608.00 (243.48)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 506.00 (120.22) | 577.77 (130.26)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 523.33 (128.55) | 592.85 (113.39)

3. Primary Outcome: Sleep Latency (SL)
Description: Sleep Latency: time taken to fall asleep, in minutes (as recorded in daily sleep diary)
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
minutes
  Baseline | 58.33 (51.01) | 47.50 (30.21)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 45.00 (41.96) | 33.33 (21.50)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 31.38 (26.98) | 41.42 (40.28)

4. Primary Outcome: Number of Awakenings
Description: As recorded in daily sleep diary
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
number of awakenings
  Baseline | 3.53 (1.84) | 3.70 (2.11)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 3.06 (1.27) | 3.11 (1.76)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 2.38 (0.78) | 3.42 (1.99)

5. Primary Outcome: Total Sleep Time (TST)
Description: minutes spent asleep as recorded in daily sleep diary
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
minutes
  Baseline | 255.66 (172.57) | 370.50 (184.98)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 339.33 (161.04) | 454.44 (178.68)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 409.44 (80.98) | 437.14 (118.73)

6. Primary Outcome: Sleep Efficiency (SE)
Description: [(TST/ TIB)X 100], (%) as recorded in daily sleep diary
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of efficient sleep
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
percentage of efficient sleep
  Baseline | 55.54 (62.44) | 62.44 (20.73)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 66.31 (24.01) | 77.48 (15.32)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 80.07 (11.65) | 75.06 (19.30)

7. Primary Outcome: Sleep Quality (SQ)
Description: As recorded in daily sleep diary. Visual analog scales (VAS) Sleep Quality Ratings 0-100, 0= extremely poor sleep quality, (shallow and unrefreshing) and 100=excellent sleep quality (deep and refreshing)
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
units on a scale
  Baseline | 44.40 (18.86) | 37.90 (13.89)
  6 week follow-up: number analyzed (Participants) | 15 | 9
  6 week follow-up | 52.46 (19.96) | 55.33 (19.93)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 59.16 (23.12) | 55.71 (11.85)

8. Primary Outcome: WASO as Assessed by Actigraphy
Description: Subjects wore a Mini Mitter Actiwatch for two continuous weeks at each assessment periods to provide an objective index compared to the assessments made by daily sleep journal. Device is lightweight and worn on non-dominant wrist and contains and omni-directional accelerometer. The accelerometer records the occurrence and degree of motion with a minimal resultant force of .01g. Data are stored as activity counts within a specified epoch. WASO recorded by device = total minutes of wakefulness after sleep onset, in minutes.
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 12
minutes
  Baseline | 64.70 (39.14) | 59.43 (15.81)
  6 week follow-up: number analyzed (Participants) | 14 | 11
  6 week follow-up | 56.30 (25.34) | 56.06 (250.80)
  12 week follow-up: number analyzed (Participants) | 11 | 9
  12 week follow-up | 59.70 (39.18) | 65.29 (17.99)

9. Primary Outcome: TST as Assessed by Actigraphy
Description: Subjects wore a Mini Mitter Actiwatch for two continuous weeks at each assessment periods to provide an objective index compared to the assessments made by daily sleep journal. Device is lightweight and worn on non-dominant wrist and contains and omni-directional accelerometer. The accelerometer records the occurrence and degree of motion with a minimal resultant force of .01g. Data are stored as activity counts within a specified epoch. TST recorded by device = total minutes spent asleep
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 12
minutes
  Baseline | 340.07 (71.23) | 367.95 (79.73)
  6 week follow-up | 337.93 (75.00) | 405.88 (79.29)
  12 week follow-up: number analyzed (Participants) | 11 | 9
  12 week follow-up | 336.84 (87.63) | 394.77 (96.86)

10. Primary Outcome: Sleep Efficiency as Assessed by Actigraphy
Description: Subjects wore a Mini Mitter Actiwatch for two continuous weeks at each assessment periods to provide an objective index compared to the assessments made by daily sleep journal. Device is lightweight and worn on non-dominant wrist and contains and omni-directional accelerometer. The accelerometer records the occurrence and degree of motion with a minimal resultant force of .01g. Data are stored as activity counts within a specified epoch. Sleep efficiency is the index of sleep percentage recorded, equal to total sleep time divided by the time in bed X 100 = X%.
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 12
percentage of time asleep
  Baseline | 73.32 (12.34) | 76.83 (8.74)
  6 week follow-up: number analyzed (Participants) | 14 | 11
  6 week follow-up | 74.77 (8.87) | 79.94 (7.49)
  12 week follow-up | 73.95 (14.15) | 75.16 (7.58)

11. Primary Outcome: Sleep Latency as Assessed by Actigraphy
Description: Subjects wore a Mini Mitter Actiwatch for two continuous weeks at each assessment periods to provide an objective index compared to the assessments made by daily sleep journal. Device is lightweight and worn on non-dominant wrist and contains and omni-directional accelerometer. The accelerometer records the occurrence and degree of motion with a minimal resultant force of .01g. Data are stored as activity counts within a specified epoch. Sleep latency is the time taken to fall asleep, or equal to lights out- sleep onset (sleep onset: time when sleep is first scored after lights out, first scorable epoch).
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 12
minutes
  Baseline | 46.25 (58.44) | 26.79 (24.73)
  6 week follow-up: number analyzed (Participants) | 14 | 11
  6 week follow-up | 39.31 (48.31) | 24.87 (17.06)
  12 week follow-up: number analyzed (Participants) | 11 | 9
  12 week follow-up | 24.71 (27.42) | 38.89 (23.49)

12. Primary Outcome: Insomnia Severity Index (ISI) Mean Total Scores
Description: The ISI is made up of 7 questions, each possible of earning a score of 0-4, making the total range 0-28, where 0 indicates no severity/no problem with sleep and therefore no insomnia, or 28, being very severe with the highest level of insomnia
Time Frame: Mean of baseline, 6 week follow-up, and 12 week follow-up
Population: Data was not included for all participants, as some were unable to complete the task.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 14 | 11
  Baseline | 15.64 (6.02) | 16.64 (4.98)
  6 week follow-up | 12.57 (4.65) | 10.71 (6.38)
  12 week follow-up: number analyzed (Participants) | 12 | 13
  12 week follow-up | 10.25 (5.19) | 13 (6.33)

13. Primary Outcome: Diffuse Noxious Inhibitory Control (DNIC) Index Scores
Description: PPTh:a somedic algometer's 1cm2 rubber probe was placed over muscle belly, with pressure increasing steadily at constant rate (30kPA/Sec), until subject indicated that s/he "first felt pain." PPTh ratings were obtained on right brachioradialis & right trapezius in a random order (average was taken from both areas at each time point). During each cold pressor task, participants immersed contralateral hand (left) up to wrist, in a circulating cold water bath maintained at 4°C. 20 seconds after commencing hand immersion, PPTh was re-assessed on either right brachioradialis or right trapezius (the same site as baseline assessment). After PPTh assessment, participants removed hands from water. DNIC was measured as the % change in PPTh during cold pressor, relative to baseline PPTh [i.e., (mean PPTh during cold pressor / mean PPTh prior to cold pressor)*100]. Increase in PPTh during cold pressor (i.e., percentage scores above 100) reflects normal functioning of pain-inhibitory processes.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of PPTh
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 13
percentage change of PPTh
  Baseline | 1.23 (0.30) | 1.19 (0.15)
  6 week follow-up: number analyzed (Participants) | 14 | 12
  6 week follow-up | 1.26 (0.31) | 1.23 (0.25)
  12 week follow-up: number analyzed (Participants) | 12 | 12
  12 week follow-up | 1.16 (0.24) | 1.14 (0.19)

14. Primary Outcome: Temporal Summation (TS)
Description: TS :maximum windup pain rating - first windup pain rating (0-100). Contact heat stimuli at non tissue damaging temperatures were delivered using computer driven, peltier-element-based stimulator (Medoc, TSA II), with a 9 cm2 probe applied to left forearm. In order to assess temporal summation, three sequences of 10 heat pulses each (with stimulus temperatures of 46 degrees C, 48 degrees C, and 50 degrees C, in random order) were applied to left dorsal forearm. The thermode remains in fixed position during administration of 10 heat pulses that constitute a sequence. Within each sequence, successive thermal pulses at a given temperature are delivered for a duration of approximately 0.5 sec each, with a 2.5-sec inter-pulse interval. The rate of rise & fall of the thermode temp. is set at the device max .of 10 degrees C / S. Subjects verbally rate the perceived intensity of each thermal pulse on a 0-100 rating scale & may terminate the procedure at any time.100=max tolerable intensity
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up at 46, 48, and 50 degrees C
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 11
units on a scale
  Baseline 46 degrees C | 9.20 (16.08) | 7.80 (12.93)
  6 week follow-up 46 degrees C: number analyzed (Participants) | 12 | 11
  6 week follow-up 46 degrees C | 6.41 (9.69) | 6.50 (7.47)
  12 week follow-up 46 degrees C: number analyzed (Participants) | 13 | 9
  12 week follow-up 46 degrees C | 5.22 (7.45) | 3.33 (7.07)
  Baseline 48 degrees C | 20.40 (41.90) | 4.72 (6.77)
  6 week follow-up 48 degrees C: number analyzed (Participants) | 12 | 9
  6 week follow-up 48 degrees C | 5.75 (8.72) | 8.11 (11.38)
  12 week follow-up 48 degrees C: number analyzed (Participants) | 13 | 9
  12 week follow-up 48 degrees C | 5.23 (8.70) | 4.55 (4.13)
  Baseline 50 degrees C: number analyzed (Participants) | 15 | 10
  Baseline 50 degrees C | 17.06 (23.09) | 21.00 (20.25)
  6 week follow-up 50 degrees C: number analyzed (Participants) | 11 | 10
  6 week follow-up 50 degrees C | 13.27 (19.66) | 18.00 (20.30)
  12 week follow-up 50 degrees C: number analyzed (Participants) | 13 | 9
  12 week follow-up 50 degrees C | 18.84 (23.82) | 20.77 (28.92)

15. Primary Outcome: Mean Level of Pain Experienced Throughout the Day
Description: Assessed using a Daily Pain Diary with a scale 0-100, 0 being no pain, 100 being the most severe/intense
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 10
units on a scale
  Baseline | 48.79 (19.63) | 52.40 (18.87)
  6 week follow-up: number analyzed (Participants) | 14 | 8
  6 week follow-up | 42.21 (18.34) | 44.43 (28.39)
  12 week follow-up: number analyzed (Participants) | 9 | 7
  12 week follow-up | 38.12 (19.11) | 42.88 (25.53)

16. Primary Outcome: Pain as Assessed by the Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) Pain Severity Subscale
Description: The WOMAC is a quality of scale life made up of three domains, pain, stiffness, and disability which each comprising of 5, 2, and 7 questions, respectively. A VAS was used for each subscale. Pain was assessed on a scale of 0-100, with 0 being absolutely no pain and 100 being maximum pain.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 12 | 11
  Baseline | 21.62 (10.75) | 24.88 (13.79)
  6 week follow-up | 19.18 (12.03) | 24.41 (13.74)
  12 week follow-up: number analyzed (Participants) | 13 | 14
  12 week follow-up | 14.85 (11.04) | 19.89 (14.15)

17. Secondary Outcome: Heat Pain Threshold
Description: Contact heat stimuli at non tissue damaging temperatures were delivered using computer driven, peltier-element-based stimulator (Medoc, TSA II), with a 9 cm2 probe applied to the left forearm. The thermode was affixed snugly via Velcro straps to ensure even skin contact and repositioned to an adjacent site after each trial to minimize sensitizationHPTh was assessed on the left ventral forearm using an ascending method of limits paradigm; from a non-painful 32°C baseline, the temperature was steadily increased at 0.5°C/sec. Two trials of heat pain threshold were conducted. Averages of both trials are presented from respective time point below. Subjects push a button when the stimulus "first feels painful" The temperature (degrees Celsius) at the time button is pushed is automatically recorded.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 14
degrees Celsius
  Baseline: number analyzed (Participants) | 15 | 13
  Baseline | 43.38 (4.71) | 42.77 (3.51)
  6 week follow-up | 43.41 (5.41) | 42.19 (3.95)
  12 week follow-up: number analyzed (Participants) | 14 | 13
  12 week follow-up | 43.31 (4.61) | 42.49 (4.38)

18. Secondary Outcome: Heat Pain Tolerance (HPTOL)
Description: Contact heat stimuli at non tissue damaging temperatures were delivered using computer driven, peltier-element-based stimulator (Medoc, TSA II), with a 9 cm2 probe applied to the left forearm. The thermode was affixed snugly via Velcro straps to ensure even skin contact and repositioned to an adjacent site after each trial to minimize sensitization. HPTOL was assessed on the left ventral forearm using an ascending method of limits paradigm; from a non-painful 32°C baseline, the temperature was steadily increased at 0.5°C/sec. Two trials of HPTOL were conducted. An average of both trials at each respective time point is presented below. Subjects push a button when the stimulus "becomes intolerable." The temperature (degrees Celsius) at the time button is pushed to terminate the stimulation is automatically recorded.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 14
degrees Celsius
  Baseline: number analyzed (Participants) | 15 | 13
  Baseline | 47.65 (2.28) | 46.56 (2.80)
  6 week follow-up | 47.54 (2.26) | 46.87 (3.56)
  12 week follow-up: number analyzed (Participants) | 14 | 13
  12 week follow-up | 47.92 (2.24) | 46.67 (3.93)

19. Secondary Outcome: Pressure Pain Threshold
Description: A Somedic algometer was used to assess pressure pain threshold (PPTh) similar to previous studies. The algometer's 1cm2 rubber probe was placed over the muscle belly, with the pressure increased steadily at a constant rate (30kPA/Sec), until the subject indicated that s/he "first felt pain." PPTh was assessed 2 times each, bilaterally, at (in a randomized order) the masseter muscle trapezius muscle, and at the proximal third of the brachioradialis muscle (forearm). The scores from each location were averaged for each participant at that respective time point. The same site was never stimulated consecutively. At least 90 s were maintained between successive stimuli
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kPA
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 15 | 14
kPA
  Baseline | 300.91 (111.13) | 267.93 (111.50)
  6 week follow-up | 322.24 (107.82) | 287.29 (107.01)
  12 week follow-up | 381.92 (199.33) | 309.15 (81.16)

20. Secondary Outcome: Quality of Life as Assessed by the Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) Disability Subscale
Description: The WOMAC is a quality of scale life made up of three domains, pain, stiffness, and disability which each comprising of 5, 2, and 7 questions, respectively. A VAS was used for each subscale. Disability was assessed on a VAS of 0-100, with 0 being absolutely no disability and 100 being maximum disability.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 12 | 11
  Baseline | 64.32 (41.26) | 74.69 (46.18)
  6 week follow-up | 62.26 (45.878) | 79.71 (47.79)
  12 week follow-up: number analyzed (Participants) | 13 | 14
  12 week follow-up | 56.13 (48.11) | 70.44 (50.75)

21. Secondary Outcome: Quality of Life as Assessed by the Short Form-36 (SF-36) Physical Health Component Summary
Description: The SF-36 is a broad, well normed measure of quality of life, comprised of 36 questions aggregated into 8 domains/dimensions. The Physical Component Summary was used here as a global index of physical health functioning. Scale 0-100, with 0 being worst functional level, 100 being the best.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 13 | 11
  Baseline | 57.61 (25.91) | 52.73 (23.38)
  6 week follow-up | 60.60 (27.48) | 49.44 (28.94)
  12 week follow-up: number analyzed (Participants) | 13 | 13
  12 week follow-up | 65.00 (21.69) | 49.40 (28.41)

22. Secondary Outcome: Quality of Life as Assessed by the Short Form-36 (SF-36) Mental Health Component Summary
Description: The SF-36 is a broad, well normed measure of quality of life, comprised of 36 questions aggregated into 8 domains/dimensions. The Mental Component Summary was used here as a global index of mental health functioning. Scale 0-100, with 0 being worst functional level, 100 being the best.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 13 | 11
  Baseline | 50.40 (9.56) | 45.78 (7.88)
  6 week follow-up | 51.68 (7.73) | 45.86 (7.06)
  12 week follow-up: number analyzed (Participants) | 13 | 13
  12 week follow-up | 50.71 (5.89) | 47.04 (11.05)

23. Secondary Outcome: Joint Stiffness as Assessed by the Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC) Joint Stiffness Subscale
Description: The WOMAC is a quality of scale life made up of three domains, pain, stiffness, and disability which each comprising of 5, 2, and 7 questions, respectively. A VAS was used for each subscale. Joint Stiffness was assessed on a VAS scale of 0-20, with 0 being no joint stiffness, and 20 being maximum stiffness.
Time Frame: Mean of baseline, 6 week follow-up and 12 week follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Eszopiclone
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline: number analyzed (Participants) | 12 | 11
  Baseline | 10.17 (5.60) | 12.86 (5.05)
  6 week follow-up | 7.55 (5.74) | 12.17 (4.41)
  12 week follow-up: number analyzed (Participants) | 13 | 14
  12 week follow-up | 6.86 (5.89) | 11.32 (5.61)

ADVERSE EVENTS:
Time Frame: Participants were followed for study duration, up to 12 weeks
Arm/Group | Placebo | Eszopiclone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 5/16 | 7/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Eszopiclone (N=14)
Restlessness, anxiety, agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Other Mild to Moderate (Not Recorded) (Product Issues) | 5 (5) | 6 (6) — It is noted that no serious adverse events (AEs) occurred. Only the number of participants who experienced mild to moderate AEs is available & has been reported. However, further information in regards to the specific AE has since been lost.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes